CLINICAL TRIAL: NCT04910997
Title: Heart Rate Variability-Guided Exercise Training in Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol closed, no participants enrolled, difficulty enrolling, funding ended.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Erin Vidra, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0165; 1-17-JDF-073 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2021-05-18; First posted 2021-06-02 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Diabetes Mellitus, Type 2; Type 2 Diabetes Mellitus in Obese
Keywords: Exercise; Aerobic exercise; Exercise training; Glucose control; Autonomic function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HRV Group (Experimental): Heart rate variability training group
  Interventions: Other: Aerobic exercise training
- Traditional Exercise Group (Active Comparator): Traditional (e.g. standard) exercise training
  Interventions: Other: Aerobic exercise training
- Control Group (No Intervention): Usual care

INTERVENTIONS:
Other: Aerobic exercise training — Combination of supervised and home-based aerobic exercise training
  Arms: HRV Group; Traditional Exercise Group

SUMMARY:
The primary aim of this randomized clinical trial is to determine the effectiveness of a 16 wk individualized aerobic exercise program, using heart rate variability to guide the exercise prescription, for increasing aerobic capacity of individuals with type 2 diabetes, compared to a traditional exercise training paradigm and usual care. To accomplish this aim the investigators plan to test for greater improvements in: 1) fitness (primary outcome); as well as secondary variables of 2) cardiovascular autonomic function via baroreflex function; 3) glucose control (HbA1c); and 4) psychosocial factors.

DETAILED DESCRIPTION:
This study will examine participant's fitness levels before and after a 16 week intervention period. There are two study visits prior to starting the intervention period. During Baseline Study Visit #1, the investigators will take a health history, determine the height and weight of the participants, and have participants complete a physical activity questionnaire and a 3-day diet log, as well as determine muscle and fat mass, followed by tests that examine how blood vessels function, and lastly a treadmill test to determine aerobic fitness. During Baseline Study Visit #2, which takes place 5-7 days later, the investigators will measure blood pressure, heart rate, and glucose control through a glucose challenge test. The glucose challenge tests requires taking ~3 Tablespoons of blood to be assessed for glucose, insulin and hemoglobin A1c. Lastly, participants will complete 3 questionnaires regarding quality of life, fatigue, and depression.

After completion of the two pre-training data collection visits, participants will be randomized to 1 of 3 groups: 1) HRV-guided exercise group (HRV); 2) traditional exercise training group (TRAD); or 3) usual care group. There will be approximately 30 subjects in each group, providing an equal chance of being assigned to either group. Both the HRV and TRAD groups will participate in a combined lab-supervised and home-based exercise program (with 1 day1 per week supervised in the laboratory and 3 days per week at home) over the course of 16 weeks. Furthermore, both exercise groups will participate in online/phone counseling in order to provide support. Specifically, participants will be provided with a phone number to the lab to call study personnel for assistance if needed. Weekly internet video chats through Zoom or phone calls, if Zoom is unavailable, will be conducted by a trained exercise-behavior change coach to help participants focus on self-efficacy, outcome expectations, impediments (barriers), and goal setting.

Post-training testing Visits #3 and #4 Visits #3 and #4 will be identical to visits #1 and 2, with the exception that the demographic questionnaire will not be administered again. This will mean there is a total of 100 mL of blood taken over the course of the entire study, between Visits 2 and 4 combined, which will total ~6 total Tablespoons.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index range = 30.0 to 40.0 kg/m2
* Being sedentary (<1 h regular physical activity/wk)
* Medication stable for 3 mo.
* Current use of physician confirmed diabetes medication, fasting glucose values ≥ 126 mg/dL and 2 hr oral glucose tolerance test (OGTT) values ≥ 200 mg/dL will be used as the criteria for type 2 diabetes

Exclusion Criteria:

* Type 1 diabetes, [insulin use]
* Major depressive disorder
* Severe neuropathy
* Current tobacco use (must have quit for 1 yr or more if a previous user)
* Renal, liver, peripheral artery, or carotid artery disease
* Current cancer (must be at least 6 mo cancer-free)
* Beta-blockers
* Perimenopausal women, post-menopausal women experiencing hot flushes and not on hormone therapy
* Alcohol consumption greater than 7 drinks/wk
* Acute coronary syndrome within the last 6 mo, heart failure, pacemaker, and any additional contraindications to participation in exercise testing or an exercise training program.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-05-02 (Estimated); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Peak aerobic capacity (fitness) | 4 months
  Aerobic capacity (e.g. fitness) will be measured during a treadmill test that assess how much oxygen the muscles need during exercise. Aerobic capacity (VO2peak) will be reported as mL/min/kg.

SECONDARY OUTCOMES:
Glucose control | 4 months
  HbA1c (glycated hemoglobin) will be the marker of glucose control in this study. HbA1c will be reported as a percentage (%).
Baroreflex sensitivity | 4 months
  This secondary outcome will be our assessment of autonomic function, whereby blood pressure and heart rate are assessed in relation to each other to create a variable called baroreflex sensitivity and reported as ms/mm Hg. Baroreflex sensitivity is defined as the change in interbeat interval (IBI) in milliseconds per unit change in BP.
Quality of life questionnaire | 4 months
  This will be assessed using the Short-Form (SF)-36 Health Survey questionnaire. Scores range between 0-100. A higher score indicates a better health status.
Fatigue severity scale | 4 months
  This outcome will assess perceived fatigue via a questionnaire that contains 9 questions. The minimum score is 9, with the maximum score being 63. The higher the score the greater the fatigue severity.
Depression questionnaire | 4 months
  This outcome will be assess via the Hospital Anxiety and Depression Scale (HADS), which is a questionnaire. There are 14 questions, and the scores can range between 0 to 21 for depression, and 0 to 21 for anxiety. A lower score means less depressive symptoms and/or anxieity.

CONTACTS AND LOCATIONS:
Overall Officials: Baynard, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No